CLINICAL TRIAL: NCT04866810
Title: The Effect of Diet and Exercise on ImmuNotherapy and the Microbiome (EDEN)
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: On hold pending planned interim analysis.
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 10000251; 000251-C
Record Dates: First submitted 2021-04-29; First posted 2021-04-30 (Actual); Last update posted 2025-10-24 (Actual); Status verified 2025-10-22

CONDITIONS: Melanoma
Keywords: Ipilimumab; Pembrolizumab; relatlimab; nivolumab; Lymphocyte activation gene 3; LAG-3; Garmin; anti PD-1/PD-L1; Acceptance and Commitment Training (ACT)
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 1 (Experimental): Intervention
  Interventions: Behavioral: Intervention Arm
- 2 (Other): Control- Standard diet and Exercise
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: Intervention Arm — High fiber, plant based diet + exercise prescription with ACT sessions
  Arms: 1
Behavioral: Control — Standard diet and exercise recommendations
  Arms: 2

SUMMARY:
Background:

The gut microbiome is made up microorganisms. These include the good and bad bacteria that live in the digestive tract. Changes in the gut microbiome have been linked to the development of cancer. Researchers want to learn more about the effects of modulating the microbiome with diet and exercise.

Objective:

To see if nutritional intake and physical activity change the gut microbiome in people with melanoma.

Eligibility:

Adults age 18 and older with previously untreated melanoma who will be getting immunotherapy treatment for their disease.

Design:

Participants will not have visits at NIH. They will have phone calls or videocalls.

Participants will be screened with a medical history and medical record review.

Participants will give stool samples. They will fill out surveys about their health, feelings, diet, and exercise.

Participants will be put in 1 of 2 groups. They will follow their group s plan for 4 months. They will be contacted throughout the study.

Intervention Group participants will follow a plant-based, high-fiber diet. They will do at least 150 minutes of moderate or 75 minutes of high-intensity exercise per week. They will have sessions with psychology staff to help them make positive lifestyle changes.

Control Group participants will be taught healthy eating and exercise guidelines. But they will not be asked to change their diet or exercise habits.

All participants will record what they eat in the MyFitnessPal app. They will get a scale to measure their weight each week. They will wear a Garmin(R) physical activity tracker at all times. They can take the tracker off to bathe or shower.

Participation will last for 6 months....

DETAILED DESCRIPTION:
Background:

The human gut microbiome is a topic of growing research interest because it modulates many systems, including immune function; and, alterations of the microbiome have been associated with the development of many diseases, including cancer.

Optimization of the gut microbiome can increase the probability of responding to immune checkpoint inhibitor therapy with responders exhibiting a higher level of gut microbial diversity than non-responders. Therefore, efforts are underway to investigate the effects of

modulating the microbiome on response to immune checkpoint inhibitor therapy.

Diet is a major modulator of the gut microbiome. In particular, a high-fiber, plant-based diet promotes greater gut microbial diversity while diets high in animal fats and protein are associated with lower gut microbial diversity.

Exercise has been shown to increase gut microbial diversity independent of diet in both mice and humans. In addition, exercise has long been known to lower cancer risk and improve outcomes in cancer patients, possibly through its ability to enhance immune

function.

Although diet and exercise prescriptions are cost-effective and implementable on a large scale, poor compliance is a major issue. Acceptance and Commitment Training (ACT) can help improve participant engagement and compliance with lifestyle change recommendations.

In melanoma participants, we hypothesize that the combination of a high-fiber, plant-based diet and exercise will increase gut microbial diversity and potentially increase the probability of responding to immune checkpoint inhibitor therapy.

Objectives:

To determine the feasibility of conducting a decentralized clinical trial involving diet and exercise prescriptions with stool sample collections in melanoma participants who will be undergoing treatment with immunotherapy.

Eligibility:

* Adults with melanoma who will be undergoing treatment with one of the following immunotherapy options: ipilimumab and nivolumab, relatlimab and nivolumab, pembrolizumab, or nivolumab.
* Adequate organ function as defined by the liver, kidney, and hematologic laboratory testing.
* Participants who have recently used antibiotics, probiotics, fiber supplements, or any other products/medications that can significantly alter the gut microbiome will be excluded.

Design:

Feasibility trial wherein participants will be randomized in a 1-to-1 fashion to the following arms:

Intervention Arm: 30 participants will be instructed to adopt a high-fiber, plant-based diet and to engage in at least 150 minutes of moderate or 75 minutes of vigorous intensity exercise per week.

Control Arm: 30 participants will be educated on general healthy eating and exercise guidelines, but they will not be instructed to change their behavior.

All participants will be asked to periodically record dietary intake (in the MyFitnessPal app or other logs, if needed), to wear a Garmin (trademark) physical activity tracker, and to collect stool samples periodically. Feasibility will be determined by assessing whether greater than or equal to 60 percent of participants in each arm adhere to their respective protocols.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Participants must have histologically or cytologically confirmed melanoma that has not been treated with any systemic therapy in the past 30 days.
* Participants must be planning to undergo immunotherapy treatment with one of the following options: ipilimumab and nivolumab, relatlimab and nivolumab, pembrolizumab, or nivolumab. Note: This treatment is permissible to have started up to 14 days prior to completion of baseline assessments on this study to still be eligible for enrollment.
* Age >= 18 years and English speaking. English-language ability is required because a portion of the study involves reading and responding to English-language questionnaires, along with creating a free response spoken answer to a question, where the information will be transcribed and analyzed.
* Willingness and capability to comply with diet and exercise prescriptions, use the MyFitnessPal app, wear the Garmin (trademark) device, complete surveys, and provide stool samples. Participants must own a smartphone capable of running the MyFitnessPal and Garmin Connect (trademark) apps.
* ECOG performance status <=2 (Karnofsky >60 percent).
* The ability of the subject to understand and the willingness to sign a written informed consent document.

EXCLUSION CRITERIA:

* Participants who are receiving any investigational agents.
* Any concurrent malignancy that requires active systemic therapy
* Any health condition that requires treatment with cytotoxic chemotherapy or targeted therapy
* Medical contraindications to the study diet and/or exercise prescriptions as determined by a physician
* Self-reported dietary and/or exercise restrictions that would preclude adherence to the study diet and exercise prescriptions
* Systemic antibiotic use within the past 30 days
* Use of probiotic supplements (probiotic foods such as yogurt, kefir, sauerkraut, etc., are permissible), fiber supplements, bile acid

sequestrants, weight loss supplements, or appetite suppressants within the last 30 days.

* Women known to be pregnant or lactating are excluded from the study because it is unknown if the study diet and exercise prescriptions may have deleterious effects on the child and/or mother in the context of pregnancy/breastfeeding.
* Current smoker or < 8 weeks since smoking cessation. There is evidence that smoking may alter the microbiome.
* Heavy drinker defined as >14 alcoholic drinks per week
* Current illicit drug use. There is evidence that illicit drug use may alter the microbiome.
* Diagnosis of diabetes mellitus type I or II that requires treatment
* Uncontrolled intercurrent illness including, but not limited to, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2023-07-25 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
feasibility of conducting a decentralized clinical trial involving diet and exercise prescriptions with stool sample collections in patients receiving immunotherapy | 43 days
  Assessing compliance with study requirements (e.g., logging diet, physical activity per the fitness tracker, completing PROs), assessed per arm; 60% compliance is a success

SECONDARY OUTCOMES:
Progression Free Survival (PFS) | through day 113
  PFS will be evaluated on the two arms using a Kaplan-Meir curve and compared using a log-rank test.
Quality of Life (QOL) | baseline, day 43 and day 113
  QOL factors in the PRO surveys will be measured using T-scores and T-tests or ANOVA.
Objective Response Rate (ORR) | through day 113
  Response rates will be compared using a one-tailed Fisher's exact test to determine if the response rate exhibits a trend toward improvement with lifestyle intervention

CONTACTS AND LOCATIONS:
Overall Officials: James L Gulley, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (2):
- United States (2):
  - Loma Linda University, Loma Linda, California
  - National Institutes of Health Clinical Center, Bethesda, Maryland

IPD SHARING:
Plan to Share IPD: Yes
All IPD recorded in the medical record will be shared with intramural investigators upon request. All IPD recorded in the medical record will be shared with intramural investigators upon request. In addition, all large scale genomic sequencing data will be shared with subscribers to dbGaP.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data available during the study and indefinitely. Genomic data are available once genomic data are uploaded per protocol GDS plan for as long as database is active
Access Criteria: Clinical data will be made available via subscription to BTRIS and with the permission of the study PI. Genomic data are made available via dbGaP through requests to the data custodians.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_000251-C.html